CLINICAL TRIAL: NCT03880201
Title: Evaluation of the Ability of Perfusion Index in Detection of Ulnar Nerve Sparing During Ultra Sound Guided Supraclavicular Block
Brief Title: Perfusion Index in Detection of Ulnar Nerve Sparing During Supraclavicular Block
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Other Study IDs: N-30-2018
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Perfusion Index as an Early Predictor of Ulnar Nerve Sparing in Supraclavicular Block; Perfusion Index as an Early Predictor of Successful Supraclavicular Block
Keywords: perfusion index.ulnar nerve sparing. supraclavicular blocK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient undergoing upper limb orthopaedic surgery: The study will be performed on patient undergoing upper limb orthopaedic surgery which will be performed under ultrasound guided supraclavicular block.
  Interventions: Procedure: ultrasound guided supraclavicular block; Device: Masimo SET pulse oximetry (Masimo Corporation, Irvine, CA, USA)

INTERVENTIONS:
Procedure: ultrasound guided supraclavicular block — The linear transducer will be applied firmly above the clavicle in the coronal oblique plane the 22-gauge needle will be inserted at the lateral side of the ultrasound probe using In-plane approach. The needle will be advanced towards the target nerves inferior, lateral and superficial to subclavian artery respectively. Local anesthetic solution is injected between 20 to 25 ml.
  Motor block will be assessed as follow Radial nerve = Push the arm by extending the forearm at the elbow against the resistance, musculocutaneous nerve = Resisting the pull of the forearm at the elbow, median nerve = Thumb and second digit pinch, ulnar nerve = Thumb and fifth digit pinch.
  Sensory block will be assessed by using piece of ice in the distribution of median, ulnar, radial and musculocutaneous nerves.
Device: Masimo SET pulse oximetry (Masimo Corporation, Irvine, CA, USA) — Masimo reading of PI values will be recorded every minute (at both index and fifth digits) for 20 minutes then every 3 minutes for 30 minutes.

SUMMARY:
The aim of this study to evaluate the ability of perfusion index to detect ulnar sparing and to estimate the proper time for the perfusion index ratio to determine successful block.

DETAILED DESCRIPTION:
On arrival to the operating room, patients will be connected to standard continuous monitoring; i.e. 5 lead electrocardiography (ECG), pulse oximetry, and automated non-invasive blood pressure monitoring (NIBP) every 5 minute. Two radical-7 (masimo set) devices will be connected the patient through two probes. The probes will be connected to both index and fifth digit to have a baseline reading before block performance. After block performance, PI will be continuously monitored for 30 minutes.

2-Anesthetic technique

Supraclavicular block:

Equipment and preparation:

* Ultrasound machine with linear transducer (8-14 MHz) (Siemens acusonx300, Korea).
* 5-cm, 22-gauge insulated block needle
* Sterile gloves, sterile sleeve, and gel (Or other coupling medium; e.g. Saline)
* 20 to 25 ml of 0.5% bupivacaine + 2% lidocaine in equal volumes

Patient position:

The block can be performed while the patient is in the supine, semi-sitting, with the Patient's head turned away from the side to be blocked with slight elevation of the head of the bed which is often more comfortable for the Patient and allows for better drainage and less prominence of the neck veins.

Technique:

After sterilization and local anaesthetic infiltration of skin, the linear transducer will be applied firmly above the clavicle in the coronal oblique plane to view the transverse section of the subclavian artery, pleura, first rib and brachial plexus (which is recognized as around or oval compact groups of hypo-echoic nerves, located lateral and superficial to the pulsatile subclavian artery and superior to the first rib). The 22-gauge needle will be inserted at the lateral side of the ultrasound probe using In-plane approach. The block needle will be advanced along the long axis of the transducer (from lateral to medial). The needle will be advanced towards the target nerves inferior, lateral and superficial to subclavian artery respectively. Local anesthetic solution is injected so as to cause hydro dissection of the planes around the plexus the volume of local Anesthetic used is usually between 20 to 25 ml.

Motor block will be assessed as inability to flex elbow and hand joints against gravity and will be tested for each nerve as follow Radial nerve = Push the arm by extending the forearm at the elbow against the resistance, musculocutaneous nerve = Resisting the pull of the forearm at the elbow, median nerve = Thumb and second digit pinch, ulnar nerve = Thumb and fifth digit pinch (15). Sensory block will be assessed by using piece of ice in the distribution of median, ulnar, radial and musculocutaneous nerves. This assessment will take place every 5 minutes till 30 minutes and the block will be considered failed if the patient reports pain at the examined dermatomes during assessment time which needs conversion to general anesthesia. If the patient reports no sensation in the whole upper limb apart from the dermatomes supplied by ulnar nerve, which is not relieved after local infiltration of skin by local anesthetic this will be considered ulnar nerve sparing.

The block assessment will be correlated with Masimo pulse oximetry readings during the first 30 minutes of the block.

Masimo reading of PI values will be recorded every minute (at both index and fifth digits) for 10 minutes then every 3 minutes for 7 readings.

Monitoring of HR, MAP and pulse oximetry will be recorded before the block and every 5 minutes for 30 minutes after the block, then every 15 minutes till the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years and weight 60-90 kg.
* ASA physical status classification I- II
* Patients scheduled for elective upper limb surgery

Exclusion Criteria:

* • upper limb ischemia

  * Diabetic neuropathy
  * Known contraindications to regional anaesthetic techniques as coagulopathy.
  * ASA physical status class III-IV.
  * Hypovolemic patients.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study will be performed on patient undergoing upper limb orthopaedic surgery which will be performed under ultrasound guided supraclavicular block.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
PI ratio in the little digit | 10 minutes after block
  PI ratio is defined as PI at 10 minutes / PI at the baseline

SECONDARY OUTCOMES:
PI ratio in the index digit | 10 minutes after block
  PI ratio is defined as PI at 10 minutes / PI at the baseline
PI values in the index digit | every minute for 20 minutes then every 3 minutes for 30 minutes
  PI values is recorded every minute for 20 minutes then every 3 minutes for 30 minutes.
PI values in the little digit | every minute for 20 minutes then every 3 minutes for 30 minutes
  PI values is recorded every minute for 20 minutes then every 3 minutes for 30 minutes.
Time needed to reach the maximum PI | every minute for 20 minutes then every 3 minutes for 30 minutes.
  PI values is recorded every minute for 20 minutes then every 3 minutes for 30 minutes.
Time needed to reach the maximum PI ratio | every minute for 20 minutes then every 3 minutes for 30 minutes.
  PI ratio is calculated as PI at each minute after block / PI at the baseline
Incidence of ulnar nerve sparing | for 30 minutes after block

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, MD, Principal Investigator — Cairo University; Bassant abdelhamid, MD, Principal Investigator — Cairo University; Mohamed Emam, Master, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith GB, Wilson GR, Curry CH, May SN, Arthurson GM, Robinson DA, Cross GD. Predicting successful brachial plexus block using changes in skin electrical resistance. Br J Anaesth. 1988 May;60(6):703-8. doi: 10.1093/bja/60.6.703. PMID 3377954
- [Background] Sorensen J, Bengtsson M, Malmqvist EL, Nilsson G, Sjoberg F. Laser Doppler perfusion imager (LDPI)--for the assessment of skin blood flow changes following sympathetic blocks. Acta Anaesthesiol Scand. 1996 Oct;40(9):1145-8. doi: 10.1111/j.1399-6576.1996.tb05578.x. PMID 8933857
- [Background] Galvin EM, Niehof S, Medina HJ, Zijlstra FJ, van Bommel J, Klein J, Verbrugge SJ. Thermographic temperature measurement compared with pinprick and cold sensation in predicting the effectiveness of regional blocks. Anesth Analg. 2006 Feb;102(2):598-604. doi: 10.1213/01.ane.0000189556.49429.16. PMID 16428569
- [Background] Goldman JM, Petterson MT, Kopotic RJ, Barker SJ. Masimo signal extraction pulse oximetry. J Clin Monit Comput. 2000;16(7):475-83. doi: 10.1023/a:1011493521730. PMID 12580205
- [Background] Kus A, Gurkan Y, Gormus SK, Solak M, Toker K. Usefulness of perfusion index to detect the effect of brachial plexus block. J Clin Monit Comput. 2013 Jun;27(3):325-8. doi: 10.1007/s10877-013-9439-4. Epub 2013 Feb 10. PMID 23397432
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539
- [Derived] Abdelhamid B, Emam M, Mostafa M, Hasanin A, Awada W, Rady A, Omar H. The ability of perfusion index to detect segmental ulnar nerve sparing after supraclavicular nerve block. J Clin Monit Comput. 2020 Dec;34(6):1185-1191. doi: 10.1007/s10877-019-00443-4. Epub 2019 Dec 9. PMID 31820214